CLINICAL TRIAL: NCT00566449
Title: A Multi-Center, Double-Blind, Placebo-Controlled, Randomized, Parallel-Group Study to Investigate the Safety and Efficacy of JNJ-31001074 in Adults With Attention-Deficit/Hyperactivity Disorder
Brief Title: A Safety and Effectiveness Study of JNJ-31001074 in Adults With Attention-Deficit/Hyperactivity Disorder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR014608; C-2007-008; NCT00767078 (obsolete NCT alias)
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; JNJ-31001074
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — bavisant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Experimental): JNJ-31001074 10 mg daily for 4 weeks
  Interventions: Drug: JNJ-31001074
- 003 (Placebo Comparator): Placebo one dose daily for 4 weeks
  Interventions: Drug: Placebo
- 002 (Experimental): JNJ-31001074 30 mg daily for 4 weeks
  Interventions: Drug: JNJ-31001074

INTERVENTIONS:
Drug: Placebo — one dose daily for 4 weeks
  Arms: 003
Drug: JNJ-31001074 — 10 mg daily for 4 weeks
  Arms: 001
Drug: JNJ-31001074 — 30 mg daily for 4 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of JNJ-31001074 compared to placebo in adults with Attention Deficit Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This study is being done to assess safety and tolerability and to explore the effectiveness of a new, experimental drug in the treatment of attention deficit hyperactivity disorder in adults. Approximately 144 adult patients with ADHD will be recruited for the study. Patients who meet study criteria will need to stop taking any ADHD medications they are currently using. They will be randomly assigned to one of 3 treatment arms; each patient has an equal chance of receiving 10 mg JNJ-31001017, 30 mg JNJ-31001074, or placebo. Placebo has no active drug. This is a blinded study, i.e. the patient, the study doctor and the study sponsor will not know what treatment the patient receives until all patients complete the study. Patients will be dispensed a bottle containing study drug for the upcoming week at 4 of the study visits. The study doctor and the sponsor will monitor the study for the occurrence of possible side effects. In addition to a screening visit, patients will return weekly for 6 additional study visits including an end of study visit and a follow-up visit. Patients will take study drug for a total of 4 weeks. After completing the study, patients may resume other ADHD medications. Medical and ADHD history, physical examination, blood pressure, heart rate, temperature, weight and ECGs will be checked periodically throughout the study. Blood samples will be taken for standard safety laboratory tests as well as for the measurement of the drug blood level. Questionnaires relating to ADHD and cognitive testing will be administered throughout the study. Each day for four weeks, patients will take orally, at least one hour before eating in the morning, 1 tablet containing either 10 mg JNJ-31001074, 30 mg JNJ-31001074 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of attention deficit hyperactivity disorder with symptoms from age 7
* In good general health
* Willing to not take any other ADHD medication or start any behaviorial modification programs during the study
* Willing to use approved birth control throughout the study and for 3 months afterwards

Exclusion Criteria:

* Any psychiatric condition including acute mood disorder, bipolar disorder, acute obsessive-compulsive disorder (OCD), anti-social personality disorder or borderline personality disorder
* Autism, asperger's syndrome, mental retardation
* Presence of motor tics, history of Tourette's syndrome or family history of Tourette's syndrome
* History of substance use/abuse disorder or eating disorder
* History of myocardial infarction, stroke, glaucoma, seizures, hypertension, heart rhythm abnormalities or color blindness
* Use of prescription medication or herbal supplements

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary study objective is to evaluate the safety and effectiveness of JNJ- 31001074 in adult patients with ADHD. | ADHD assessments, vital signs, laboratory tests and ECGs will be collected 7 times during the study; at screening, baseline and 5 weekly visit. Adverse events will be collected throughout the study.

SECONDARY OUTCOMES:
The secondary study objective is to assess drug levels in adults with ADHD after taking JNJ-31001074. | Samples to measure drug levels in the blood will be collected three times at baseline and termination visits and once at visits done at Weeks 1, 2, and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA; Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (21):
- United States (21):
  - Irvine, California
  - Lafayette, California
  - San Francisco, California
  - Bradenton, Florida
  - Fort Myers, Florida
  - Orlando, Florida
  - South Miami, Florida
  - Eagle, Idaho
  - Libertyville, Illinois
  - Overland Park, Kansas
  - Boston, Massachusetts
  - Farmington, Michigan
  - Chapel Hll, North Carolina
  - Raleigh, North Carolina
  - Dayton, Ohio
  - Portland, Oregon
  - Media, Pennsylvania
  - Austin, Texas
  - Houston, Texas
  - Herndon, Virginia
  - Seattle, Washington